CLINICAL TRIAL: NCT03292822
Title: Apoptotic and Anti-Proliferative Effects of Licorice Extract (Licochalcone A) and Paclitaxel Chemotherapy on Human Oral Squamous Cell Carcinoma Cell Line
Brief Title: Effects of (Licochalcone A) and Paclitaxel on Human Oral Squamous Cell Carcinoma Cell Line
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Moahmed Osama mostafa, teaching assistant, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2017-09-26
Record Dates: First submitted 2017-09-12; First posted 2017-09-26 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — licochalcone A; Paclitaxel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Licochalcone A (Experimental): Licochalcone A is a chalconoid, a type of natural phenols. It can be isolated from root of Glycyrrhiza glabra (liquorice) or Glycyrrhiza inflata. It shows antimalarial, anticancer, antibacterial and antiviral (specifically against influenza neuraminidase) properties.
  Interventions: Dietary Supplement: Licochalcone A
- Paclitaxel (Active Comparator): chemotherapeutic drug
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Dietary Supplement: Licochalcone A — Licochalcone A is a chalconoid, a type of natural phenols. It can be isolated from root of Glycyrrhiza glabra (liquorice) or Glycyrrhiza inflata. It shows antimalarial, anticancer, antibacterial and antiviral (specifically against influenza neuraminidase) properties in vitro.
  Arms: Licochalcone A
Drug: Paclitaxel — chemotherapeutic drug
  Other Names: taxol
  Arms: Paclitaxel

SUMMARY:
Oral squamous cell carcinoma (OSCC) are considered as a one of the most malignant cancers. It has prognosis due to its distant metastasis and obvious destruction which lead to low survival rate.

The conventional treatment modalities such as surgery, radiotherapy and chemotherapy are only the suitable strategies until now. Investigators cannot ignore the serious side effects of chemotherapy such as gastrointestinal upset, bone marrow suppression which cannot be overcome. For all these complications, there is a great need and demand to discover a new agents and strategies for treating OSCC.

Licorice extract, especially Licochalcone A, is one of many natural extracts that have used as a traditional in treatment of inflammation, microbial infections. Regarding antitumor effect, Licochalcone A reveals interesting results in programmed cell death and apoptosis in cancer cells such as prostate, bladder, colon and gastric cancer.

DETAILED DESCRIPTION:
Oral squamous cell carcinoma (OSCC) is considered the most common human body malignant tumor. It has poor prognosis regarding its distant lymph node metastasis and local destruction which lead to low survival rate.

Paclitaxel is a chemotherapeutic drug of the taxols group that is used in the treatment of lung, ovarian and prostate cancer. It is also used to treat breast, head and neck cancer as well as sarcoma and leukemia. Recent studies and researches explored that Paclitaxel has an important role in mitotic arrest activation and induction, which subsequently lead to cell death.

The conventional treatment strategies such as surgery, radiotherapy and chemotherapy come with low levels of expectations regarding prognosis and survival rate. On the other hand, serious side effects of chemotherapy such as renal toxicity, gastrointestinal upset and bone marrow suppression remain hazards which cannot be avoided.Thus, there is a great need to discover new agents and strategies for treating OSCC or even enhancing the effect of chemotherapy in order to reduce the dose given.

Licorice extract, Licochalcone A, is one of many natural extracts of Glycyrrhiza inflata plant. It has been used in treatment of inflammation, infections and cancer.

ELIGIBILITY:
Inclusion Criteria:

1. All head and neck squamous cell carcinoma cell lines
2. Licochalcone extracts
3. Taxols group of chemotherapy

Exclusion Criteria:

1. Animal experimental studies
2. Any cancer cell line other than squamous cell carcinoma cell lines.
3. Any chemotherapeutics other than Taxols group.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Apoptosis | 3 days
  programmed cell death

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed H El-Khadem, Phd, Study Chair — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

REFERENCES:
- [Background] Park MR, Kim SG, Cho IA, Oh D, Kang KR, Lee SY, Moon SM, Cho SS, Yoon G, Kim CS, Oh JS, You JS, Kim DK, Seo YS, Im HJ, Kim JS. Licochalcone-A induces intrinsic and extrinsic apoptosis via ERK1/2 and p38 phosphorylation-mediated TRAIL expression in head and neck squamous carcinoma FaDu cells. Food Chem Toxicol. 2015 Mar;77:34-43. doi: 10.1016/j.fct.2014.12.013. Epub 2015 Jan 5. PMID 25572524

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-22): https://cdn.clinicaltrials.gov/large-docs/22/NCT03292822/Prot_SAP_000.pdf